CLINICAL TRIAL: NCT06619574
Title: Improving TMJ Joint Positioning and Accuracy With Therapeutic Splint Fabrication Using a Dental Compass While Reducing Radiation Exposure: A Cohort Comparison
Brief Title: Temporomandibular Joint (TMJ) Positioning Accuracy and Efficiency Using a Dental Compass.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Collaborators: Lourens A. Du Preez (Unknown)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Principal Investigator, Dr. Dean Reeves Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dental Compass - 01
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Joint Syndrome
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Intervention Model Description: Cohort comparison study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Analysis Group (Experimental): Compass Use
  Interventions: Device: 3D Analysis Group
- Manual Analysis Cohort (Active Comparator): Manual Use only
  Interventions: Other: Manual Analysis Cohort

INTERVENTIONS:
Device: 3D Analysis Group — Dental Compass and Dental Compass software used for therapeutic splint fabrication
  Arms: 3D Analysis Group
Other: Manual Analysis Cohort — Manual methods used for therapeutic splint fabrication
  Arms: Manual Analysis Cohort

SUMMARY:
This study is being performed to determine if the use of the Dental Compass Articular and its software will produce therapeutic splints for TMD accurately and successfully, compare favorably with a cohort treated without the Dental Compass (for number of visits, splint modifications, and required CBCTs).

DETAILED DESCRIPTION:
Standard practice in the treatment of temporomandibular dysfunction (TMD) currently involves non-radiographically-assisted manual repositioning of the jaw followed by either an in-office cone beam computerized tomography (CBCT) or tomographic X-ray of both TMJs, and further adjustment as necessary to improve the initial bite impression.[15] At follow up visits the therapeutic splint is modified in stages to "walk" the condyle progressively into the ideal position, such as altering side shift, lateral deviation, and rotation. During this process multiple CBCTs or tomographic X-rays, and multiple direct dentist interventions, are required to find the precise joint position, involving significant radiation exposure, and significant chair time for the dentist

The key advantage of using the Dental Compass Articulator in conjunction with its software, is to identify and suggest corrections for the range of orthopedic imbalances present. Software-facilitated identification of imbalances is coupled with manipulation of yaw (anterior, posterior, lateral, or rotational movement of the mandible in a horizontal plane), pitch (rotation of the mandible in a frontal vertical plane), and roll (rotation of the mandible in a lateral vertical plane) to achieve optimal condylar and mandibular position for splint manufacture.

The goals of this study are to:

1. Determine if the use of the Dental Compass Articular and its software will produce therapeutic splints for TMD accurately and successfully, and will compare favorably with a cohort treated without the Dental Compass (for number of visits, splint modifications, and required CBCTs), and
2. Confirm a clinically important reduction in airway constriction and improvement in airway volume with us of the therapeutic splint.

ELIGIBILITY:
Inclusion Criteria for prospective active participants:

* TMJ dysfunction and pain
* CBCT indicates a non-Gelb 4/7 position or < 1.8 mm bone to bone interval between the mandibular condyle and mandibular fossa anteriorly or posteriorly.

Exclusion Criteria:

* Planning a move within 9 months.
* Unwilling to provide two phone numbers and two email contacts.
* Not willing to express a willingness to come in for 4-6 month follow up if they have marked improvement or improvement in symptoms.
* Not living within 90-minute drive from clinic
* Transportation not reliable
* Involved in any other TMD study
* Life threatening illness or major surgery planned
* Other major life stress that might interfere with completing the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of clinic visits | 3-6 months
  Number of clinic visits from initial evaluation to confirmation of final therapeutic splint provision
Number of cone beam CTs (CBCTs) | 3-6 months
  Number of CBCTs obtained from initial evaluation to confirmation of final therapeutic splint provision
Number of splint modifications | 3-6 months
  Number of splint modifications obtained from initial evaluation to confirmation of final therapeutic splint provision

SECONDARY OUTCOMES:
Gelb 4/7 position achieved during treatment (3D group only) | 3-6 months
  Yes or no for Gelb 4/7 position
Anterior joint space of 1.8 mm or more achieved during treatment (3D group only) | 3-6 months
  Yes or no for anterior joint space of 1.8 mm or more
Posterior joint space of 1.8 mm or more achieved during treatment (3D group only) | 3-6 months
  Yes or no for posterior joint space of 1.8 mm or more
Improvement in total airway volume | 3-6 months
  Change in total airway volume from use of TMJ splint
Improvement in minimum airway diameter | 3-6 months
  Change in total airway volume from use of TMJ splint

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, MD, Principal Investigator — K. Dean Reeves, M.D., P.A.
Locations (1):
- Skalff Dental Studio and Technologies 103 C West Broadway Street #3736, Gainesville, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All non identifying data
Supporting Information: Study Protocol, SAP
Time Frame: Indefinitely
Access Criteria: By email request to P.I. at DeanReevesMD@gmail.com